CLINICAL TRIAL: NCT06162364
Title: Investigation of The Effect Of Scenario-Based Three-Dimensional Video Education Utilizing Virtual Reality Glasses on Nursing Students' Surgical Handwashing and Sterile Dressing Skills
Brief Title: Surgical Hand Washing and Sterile Dressing Training With Virtual Reality Glasses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Songul Gungor, Phd Lecturer, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OsmaniyeKAUU
Record Dates: First submitted 2023-09-26; First posted 2023-12-08 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Virtual Reality
Keywords: Virtual reality; surgical nursing education; surgical handwashing and sterile dressing skills; three-dimensional video education; scenario-based training
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Intervention Model Description: A sample of 79 voluntary students was divided into three groups through simple randomization: VR group (N=27), theoretical education group (N=27), and video education group (N=25). The VR group received education using VR goggles, the theoretical group underwent traditional theoretical education, and the video group was educated through video content on surgical handwashing and sterile dressing. For the VR group, 3D videos were presented using VR goggles, while the video group experienced 2D video content. The theoretical group was allocated self-study time. Subsequent to the educational interventions, student performance, self-confidence, and satisfaction were evaluated. Data collection involved various forms assessing skills, knowledge, technology usage, method satisfaction, and self-confidence.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR group (Experimental): In this group, students were taught surgical hand washing and sterile dressing skills through theoretical training, demonstration, and VR glasses. Later, a theoretical knowledge assessment test was administered, and they were subjected to a skill evaluation exam in the laboratory.
  Interventions: Other: VR; Other: theoretical training
- theoretical training group (No Intervention): In this group, students were taught surgical hand washing and sterile dressing skills through theoretical training and demonstration. Later, a theoretical knowledge assessment test was administered, and they were subjected to a skill evaluation exam in the laboratory.
- video training group (Experimental): In this group, students were taught surgical hand washing and sterile dressing skills through theoretical training, demonstration, and two-dimensional video. Later, a theoretical knowledge assessment test was administered, and they were subjected to a skill evaluation exam in the laboratory.
  Interventions: Other: VR; Other: training with video

INTERVENTIONS:
Other: VR — playing a video using VR
  Arms: VR group; video training group
Other: theoretical training — Training was provided through theoretical education
  Arms: VR group
Other: training with video — Training was given with two-dimensional video
  Arms: video training group

SUMMARY:
ABSTRACT This study is a comparison of the impact of virtual reality on surgical handwashing and sterile dressing knowledge, skills, satisfaction, and confidence in nursing students enrolled in surgical nursing, as opposed to conventional teaching methods.

Keywords: Virtual reality, surgical nursing education, surgical handwashing and sterile dressing skills, scenario-based education, three-dimensional video education.

DETAILED DESCRIPTION:
This research is a randomized controlled experimental study aiming to investigate the impact of scenario-based three-dimensional video education using virtual reality goggles on surgical handwashing and sterile dressing skills. Volunteer nursing students, forming the research sample, were divided into three groups using a simple random sampling method. The first group was provided with an 11-minute VR experience using virtual reality goggles, repeated three times. The second group received theoretical training methods, with a one-time 30-minute session and a demonstration, followed by free study time. The third group received training three times with an 11-minute video. Three weeks later, the students' skills were assessed using a validated skills assessment form. Their confidence and satisfaction levels were evaluated through a questionnaire.

ELIGIBILITY:
Inclusion Criteria:

To be 18 years and older,

Being an active student of the Nursing Department,

Being enrolled in the Surgical Nursing Diseases Course for the first time,

Not having claustrophobia,

Not having head or neck disorders that would prevent wearing virtual reality goggles.

Exclusion Criteria:

Being a graduate of a Health Vocational High School,

Being a graduate of a pre-license health services vocational college,

Having attended any webinar, congress, or meeting related to surgical hand washing and sterile dressing,

Having professional working experience in the nursing/healthcare field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of voluntary participants | at study 1 day visit
  Researchers determined feasibility by measuring the percentage of participants who volunteered to participate and met the research criteria.

SECONDARY OUTCOMES:
Skill acquisition | at study three weeks visit.
  Researchers measured the impact of the teaching method on skill acquisition in all students using a 39-item skill assessment form.
Knowledge acquisition | at study three weeks visit
  Researchers measured the impact of the teaching method on knowledge acquisition in all students using a 10-item knowledge assessment form.
Satisfaction with VR experience | at study three weeks visit
  Researchers used a 10-point measurement form to assess the perceived change impression in students after the VR experience.
Gain in self-confidence | at study three weeks
  Researchers used a 10-point measurement form to assess the impact of the teaching method on self-confidence gain in all students.

CONTACTS AND LOCATIONS:
Locations (1):
- Songül GÜNGÖR, Merkez, Osmani̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Vrillon A, Gonzales-Marabal L, Ceccaldi PF, Plaisance P, Desrentes E, Paquet C, et al. Using virtual reality in lumbar puncture training improves students learning experience. BMC Med Educ.2022;22(1):1-8 — https://doi.org/10.1186/s12909-022-03317-7
- See also: Shin S, Park JH, Kim JH. Effectiveness of patient simulation in nursing education: Meta-analysis. Nurse Educ Today.2015;35(1):176-82 — http://dx.doi.org/10.1016/j.nedt.2014.09.009
- See also: Chen FQ, Leng YF, Ge JF, Wang DW, Li C, Chen B, et al. Effectiveness of virtual reality in nursing education: Meta-analysis. J Med Internet Res. 2020;22(9):e18290 — https://doi.org/10.2196/18290
- See also: Fleming SE, Reynolds J, Wallace B. Lights... camera... action! a guide for creating a DVD/video. Nurse Educ. 2009;34(3):118-21. — https://doi.org/10.1097/NNE.0b013e3181a0270e
- See also: Sen S, Usta E, Bozdemir H. The effect of mobile virtual reality on operating room nursing education. Teach Learn Nurs. 2022;17(2):199-202. — https://doi.org/10.1016/j.teln.2022.01.008